CLINICAL TRIAL: NCT00884039
Title: Compassionate Use of Anecortave Acetate: Clinical Protocol for the Treatment of Corticosteroid-induced Intraocular Pressure (IOP) Increases After Corneal Transplantation
Brief Title: Anecortave Acetate Injection to Treat Steroid-responsive Intraocular Pressure Increase in Cornea Transplant Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary data analysis showed insufficient efficacy to justify continuation.
Sponsor: Cornea Research Foundation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-12
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Transplant; Intraocular Pressure
Keywords: cornea; transplant; intraocular pressure; steroid response
MeSH Terms: conditions — Corneal Diseases | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 mg anecortave acetate (Active Comparator)
  Interventions: Drug: 30 mg anecortave acetate
- 15 mg anecortave acetate (Active Comparator)
  Interventions: Drug: anecortave acetate

INTERVENTIONS:
Drug: anecortave acetate — anterior juxtascleral depot of 15 mg anecortave acetate
  Arms: 15 mg anecortave acetate
Drug: 30 mg anecortave acetate — anterior juxtascleral depot of 30mg anecortave acetate
  Arms: 30 mg anecortave acetate

SUMMARY:
This study will investigate the use of anecortave acetate injection to reduce intraocular pressure (IOP) in corneal transplant recipients who are experiencing steroid-associated pressure control problems. Alternative methods of IOP control have been shown to entail serious risks. For example, reduction of topical steroids increases the risk of graft rejection, and use of glaucoma medications or glaucoma surgery increases the risk of graft failure. This study is designed to have sufficient power to detect whether a single injection can induce a clinically significant IOP reduction.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* corneal transplant recipient with intraocular pressure (IOP) greater than 24 mmHg and with relative increase in IOP of at least 10 mmHg over the pre-graft baseline

Exclusion Criteria:

* not pregnant or lactating
* intraocular surgery in the study eye within 30 days before enrolling in the study
* use of any investigational drug or treatment within 30 days before receipt of study medication
* clinical evidence of scleral thinning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W. Price, Jr., MD, Principal Investigator — Cornea Research Foundation of America
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 30 mg Anecortave Acetate | 15 mg Anecortave Acetate
Started | 5 | 2
Completed | 3 | 1
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 30 mg Anecortave Acetate | 15 mg Anecortave Acetate | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (19) | 70 (2) | 65 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure Within Normal Limits (<24 mm Hg)
Description: Intraocular pressure was measured by Goldmann applanation tonometry.
Time Frame: 1 month
Population: Per protocol
Measure: Number; unit: Participants
Arm/Group | 30 mg Anecortave Acetate | 15 mg Anecortave Acetate
Number analyzed (Participants) | 5 | 2
Participants | 2 | 1
Statistical Analysis 1: Comparison: 30 mg Anecortave Acetate vs 15 mg Anecortave Acetate; Test type: Superiority or Other; p = 0.57, Fisher Exact

ADVERSE EVENTS:
Arm/Group | 30 mg Anecortave Acetate | 15 mg Anecortave Acetate
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 4/5 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg Anecortave Acetate (N=5) | 15 mg Anecortave Acetate (N=2)
Intraocular pressure elevation (Eye disorders) | 4 (5) | 2 (3)
Eye discomfort (Eye disorders) | 1 (1) | 1 (1)
Cornea transplant rejection episode (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No